CLINICAL TRIAL: NCT04989205
Title: Examining a Community Based Intervention for Cannabis Smoking Cessation in Norway - an Observational Study
Brief Title: Community Based Cannabis Cessation Program
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: City of Oslo (Unknown); Municipality of Kristiansand (Unknown); Norway Centre for Addiction Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 005004
Record Dates: First submitted 2021-07-12; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Cannabis Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HAP - group: The target group was individuals who engaged in regular or daily cannabis use, and who were motivated to quit cannabis. The formal inclusion criteria was a Severity of Dependence Scale (SDS) score ≥4 and being ≥16 years old. Exclusion criteria was polydrug use where cannabis was not the predominating substance of use and psychiatric comorbidity that was perceived as too severe to handle at the community-based centers .
  Interventions: Behavioral: Cannabis cessation Program

INTERVENTIONS:
Behavioral: Cannabis cessation Program — Lundqvist and Ericsson developed the 'Cannabis Cessation Program' (CCP, Nordic abbreviation: HAP) in Sweden in the 1990s. The method uses a combination of cognitive therapy and psychoeducation and covers the normal withdrawal period for cannabis smoking cessation (up to 8 weeks), comprising ~15 individual sessions. It describes a medical, a psychological, and a social phase, in which the participant is helped to recognize and address typical problems related to each phase, e.g., physical and psychological withdrawal problems. The overarching aim of the program is to help cannabis users to reorganize thinking patterns that developed while they were using cannabis and increase their social and psychological coping skills in relation to quitting cannabis use. The CCP manual has been translated into eight languages, e.g., Norwegian.

SUMMARY:
The study examined a community based cannabis cessation program in Norway (CCP). The CCP uses a combination of cognitive therapy and psychoeducation and covers the normal withdrawal period for cannabis smoking cessation (up to 8 weeks), comprising ~15 individual sessions. From 2005 onwards, the CCP was implemented as a low-threshold community-based program in several Norwegian municipalities, e.g., Kristiansand, Fredrikstad and Oslo. The study had an observational one-group pre- / post test design. Outcomes was changes in cannabis use, mental distress, well-being, social network and sense of coherence (SoC) measured post-intervention (T2) and at a 3 months follow-up (T3).

ELIGIBILITY:
Inclusion Criteria:

* Severity of Dependence Scale (SDS) score ≥4

Exclusion Criteria:

* polydrug use where cannabis was not the predominating substance of use
* psychiatric comorbidity that was perceived as too severe to handle at the community-based centers

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The target group was individuals who engaged in regular or daily cannabis use, and who were motivated to quit cannabis.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-06-02 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Cannabis use | Changes from baseline to post-treatment and follow-up, on average 5 months
  Days with cannabis use last 30 days

SECONDARY OUTCOMES:
Mental distress | Changes from baseline to post-treatment and follow-up, on average 5 months
  The Hopkins Symptom Checklist (HSCL) 25-item version was used to measure mental distress. Each of the 25 items was scored on a 4-point scale (1-4). An average score was computed, indicating a global severity index of mental distress (GSI), where higher scores indicated greater distress. Clinical cut-off = 1.75
Well-being | Changes from baseline to post-treatment and follow-up, on average 5 months
  The Outcome Rating Scale (ORS) was used to assess well-being. The scale has four visual analogue items on personal, interpersonal, social, and general well-being, and each item are scored from 0 = bad up to 10 = good. The items are then summed (range 0-40) and a score <25 indicated scores expected in a clinical population.
Social network | Changes from baseline to post-treatment and follow-up, on average 5 months
  Number of current friends with and without problematic substance use
Sense of Coherence (SoC) | Changes from baseline to post-treatment and follow-up, on average 5 months
  The Sense of Coherence questionnaire, 29 item version, measures the degree to which the subject feels that he or she has a sense of control over their own lives (manageability - 10 items), that life has meaning (8 items) and that their social life is understandable (comprehensibility - 11 items). Responses to items are scored on a seven-point semantic differential scale. Scores are summed (ranges from 29 - 203) and higher scores indicated a stronger SoC

CONTACTS AND LOCATIONS:
Overall Officials: John-Kåre Vederhus, PhD, Principal Investigator — Addiction Unit, Sørlandet Hospital, Kristiansand
Locations (3):
- Norway (3):
  - Social Services, Fredrikstad Municipality, Fredrikstad
  - Kristiansand Municipality, Cannabis Cessation Program, Kristiansand
  - City Centre Outreach Service, Agency for Social and Welfare Services, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared upon request. Anonymous data will be shared upon reasonable request
Supporting Information: Study Protocol
Time Frame: Upon request
Access Criteria: Upon request

REFERENCES:
- [Derived] Vederhus JK, Rorendal M, Skardal M, Naess MO, Clausen T, Kristensen O. Successful outcomes with low-threshold intervention for cannabis use disorders in Norway - an observational study. PLoS One. 2022 Jun 16;17(6):e0269988. doi: 10.1371/journal.pone.0269988. eCollection 2022. PMID 35709178